CLINICAL TRIAL: NCT00941226
Title: Evaluation of the Quality of Life of Cerebral Palsy Child Carers
Brief Title: The Quality Of Life Of Cerebral Palsy Child Carers
Status: Completed | Type: Observational
Sponsor: Centro de Estudos Superiores de Maceio (Other)
Responsible Party: Thâmara Camylla Ribeiro de Barros Calado, Centro de Estudos Superiores de Maceió - CESMAC.
Other Study IDs: 340/07
Record Dates: First submitted 2009-07-16; First posted 2009-07-17 (Estimated); Last update posted 2009-07-20 (Estimated); Status verified 2009-07

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Caregivers; Quality of Life
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cerebral Palsy: Those kids who have cerebral palsy and are helped by carers

SUMMARY:
Cerebral Palsy (CP) is characterized by a sensory-motor deficiency, involving disturbance of muscle tone, posture and voluntary movement. Children who are afflicted need special intense care for their carers

DETAILED DESCRIPTION:
INTRODUCTION: Cerebral Palsy (CP) is characterized by a sensory-motor deficiency, involving disturbance of muscle tone, posture and voluntary movement. Children who are afflicted need special intense care for their carers. OBJECTIVE: The objective of this study was to analyze the quality of life of CP child carers attended in the physiotherapy sector of a philanthropic institution on Maceió - AL. METHODS: 62 carers were assessed in the period from the 18th to the 29th of February 2008, in which 96.7% were female carers and 3.7% male. The form for the collection of data from the carers, elaborated by the researchers and the WHOQOL-26 quality of life questionnaire were utilized as as instruments.

ELIGIBILITY:
Inclusion Criteria:

* Children who were attended by Associação dos Pais e Amigos dos Excepcionais (APAE), Maceió, Alagoas
* They had cerebral palsy

Exclusion Criteria:

* Child who had not cerebral palsy
* Child under 2 years old

Min Age: 2 Years | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CP child carers attended in the physiotherapy sector of a philanthropic institution on Maceió - AL
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2007-10; Primary Completion 2008-03 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thâmara C. R. B. Calado, Graduated, Principal Investigator — Centro de Estudos Superiores de Maceio